CLINICAL TRIAL: NCT06688591
Title: Effectiveness of an Evidence-based Multi-component Intervention Programme to Reduce Medication-related Problems Among Polymedicated Home-dwelling Older Adults: Protocol for a Multi-site Pilot Study of the OptiMed Clinical Trial
Brief Title: Protocol for a Multi-site Pilot Study of the OptiMed Clinical Trial
Acronym: OptiMed
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in finding participants for the various stages of the study
Sponsor: HES-SO Valais-Wallis (Other)
Collaborators: Polytechnic of Leiria (Unknown); Institute for Primary Health Care BIHAM, University of Bern (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 105 995
Record Dates: First submitted 2021-11-19; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Polypharmacy; Multiple Chronic Conditions
Keywords: protocol; pilot study; feasibility; informal caregivers; interprofessional collaboration; patient-centred care; medication management; home-dwelling older adults; medication safety; medication-related problems
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: The pilot OptiMed randomised pragmatic trial will focus on the feasibility components using an open-label design where participants know what they are signing up for. It will support the development of a standardised, evidence-based, multi-component, interprofessional intervention programme to reduce MRPs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Medication-management intervention programme to reduce the risks of MRPs (Experimental): The research nurse will help the older participant and their informal caregiver to implement their target education plan (t2) aimed at empowering their medication management and promoting their active engagement in reducing the risks of MRPs
  Interventions: Other: Intervention programme to optimise medication management and prevent MRPs

INTERVENTIONS:
Other: Intervention programme to optimise medication management and prevent MRPs — The intervention is based on a four-step patient empowerment process: 1) the patient understands their role; 2) the patient acquires sufficient knowledge to be able to engage with their healthcare professionals; 3) the patient improves their skills; and 4) there is a facilitating environment (30). Each older adult participant's plan will be unique and consider their preferences, medication literacy and treatment adherence.
  Other Names: Preventive intervention

SUMMARY:
Background: Optimal medication management is one of the essential preconditions for polymedicated home-dwelling older adults with multiple chronic conditions to remain at home and preserve their quality of life and autonomy. This study aims to explore the feasibility and acceptability of an evidence-based, multi-component, interprofessional intervention programme supported by informal caregivers to decrease medication related problems (MRPs) among polymedicated, home-dwelling older adults with multiple chronic conditions.

Methods: The pragmatic multi-site OptiMed pilot study will use an open-label design, where participants know what they are signing up for and will take place in primary healthcare settings in Portugal and Switzerland. The research population will comprise polymedicated home-dwelling adults aged 65 years old or more, at risk of MRPs and receiving community-based healthcare.

Discussion: This pilot study will focus on the recruitment and collaboration of study participants and piloting the feasibility of the evidence-based, multi-component, interprofessional intervention programme. The full-scale study, following on from the OptiMed pilot study, will support the development of a standardised, evidence-based, multi-component, interprofessional intervention programme to reduce MRPs. It will also be an essential part of follow-up research programmes on the multiple roles of informal caregivers, as it will put their coordination tasks into perspective with their own needs.

DETAILED DESCRIPTION:
The pilot study's primary objective is to explore the feasibility and acceptability of an evidence-based, multi-component, interprofessional intervention programme, supported by informal caregivers, to decrease MRPs among polymedicated, home-dwelling older adults with multiple chronic conditions. The pilot study will gather information about the feasibility and acceptability of recruitment, participant retention, adherence, fidelity, acceptability and satisfaction, intervention dose, and the intervention programme's overall credibility. The secondary objective is to test the different data collection tools planned for use in the full study.

After the older participant has been recruited via their nurse primary-care manager, working for their primary healthcare centre (PHC), the intervention's first component (t0) involves a baseline assessment of them at a meeting conducted by a research nurse. The research is explained to the older participant in detail, both orally and in writing, and the consent form is signed. Following this, the older participant is asked to answer some sociodemographic and health-related questions and provide a complete list of their current medication prescription. The research nurse completes a questionnaire on the risk of MRPs-doMESTIC risk. A first meeting also takes place individually with the family caregiver (who will also answer some sociodemographic and health-related questions and describe their role in medication management). The older participant is asked to identify the healthcare professional(s) (GP or specialist, nurse primary-care manager and/or community pharmacist) most involved in their medication management.

The second component (t1) involves a review of the prescribed medications in week 1, including a medication reconciliation and a structured medication analysis by the pharmacist study partner, to identify drugs with a high risk of MRPs among older adults. This will use the STOPP/START criteria, and undertreated indications or missed therapies will use the START criteria. The older adult's physician will be invited to participate in the review of prescribed medications in collaboration with the pharmacist study partner. They will discuss validated, evidence-based, internationally recognised guidelines to reconsider beneficial or non-beneficial therapies or to simplify and focus on specific care goals and adjust medications to be consistent with guidelines. If the older adult's physician adopts no changes despite the medication review (t1) highlighting their relevance, the research team will inform the older adult of their physician's decision and will invite them to proceed with the study.

Based on the baseline assessment (t0), the research nurse will use a joint consultation in week 2 to explore the needs and care goals of the older participant and their informal caregiver so as to reduce the risk of MRPs (t2). The research nurse will then design a target education plan-in collaboration with the designated healthcare professional(s)-to empower the older adult's medication management and reduce the risk of MRPs (t2). This is based on a four-step patient empowerment process: 1) the patient understands their role; 2) the patient acquires sufficient knowledge to be able to engage with their healthcare professionals; 3) the patient improves their skills; and 4) there is a facilitating environment. Each older adult participant's plan will be unique and consider their preferences, medication literacy and treatment adherence.

During weeks 3 and 4 (t3), the research nurse will help the older participant and their informal caregiver to implement their target education plan (t2) aimed at empowering their medication management and promoting their active engagement in reducing the risks of MRPs. Two joint consultations will be organised between the older adult, their informal caregiver and the research nurse (once each week). During planned home visits, the nurse will periodically evaluate older adults' medication status (primary and secondary outcomes) and promote communication between the different professional and non-professional actors involved in medication management.

The research nurse will carry out a final assessment (t4) of each older adult's risks of MRPs in week 5 (35-40 days after t0) in collaboration with the study partner pharmacist. The occurrence of MRPs and medication-related hospital admissions will be investigated. Finally, the acceptability of the interprofessional intervention programme to reduce MRPs will be assessed by the healthcare professionals designated by the older adult in a final questionnaire.

As already described, the medication-management intervention programme guiding OptiMed's pilot study comprises four components based on concurrent interacting processes previously identified by Boult and Wieland. The pilot study will explore possible biases so that they can be correctly addressed in the full study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older for both men and women
* Suffering from multiple chronic conditions (two or more)
* Managing at least four prescribed medications daily for more than 90 days (2) (explored during recruitment)
* At risk of MRPs identified using the doMESTIC RISK tool
* Living alone or with a partner, in a rural or urban area
* Supported by a Primary Healthcare Centre
* An informal caregiver is involved in medication management
* Gives written informed consent

Exclusion Criteria:

* Unable to speak and understand French
* Moderate or severe dementia criteria (≥ 10 on the Six-item Cognitive Impairment Test, 6-CIT)
* No risk of MRPs (doMESTIC RISK tool score < 5)
* No informal caregiver

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Target population is recruited | 6 months
  Number screened per month; number enrolled per month; average time delay from screening to enrolment
Study participants are retained | 6 months
  Treatment-specific retention rates (%) for study measurements (eligible / recruted / completed); reasons for drop-outs
Study participants adhere to their instructions | 6 months
  Treatment-specific rates (%) of adherence to study protocol (in-person session attendance, homework, home sessions, etc.); treatment-specific measurements of competencies
Medication review is successful | 6 months
  Treatment-specific fidelity rates in %; time invested in hours; number of discrepancies between professional sources; number of discrepancies between patient-reported medication use and professional sources n= or %; number of questions; number of items needing clarification; number of recommendations made by the pharmacist; number of pharmacist's recommendations adopted by the physician
Assessments are not considered too burdensome | 6 months
  Proportion of planned assessments that are completed (%); duration of assessment visits (minutes); reasons for drop-outs (listing); ease of use of doMESTIC RISK tool (self-reporting closed questionnaire); ease of use of structured medication review template (self-reporting closed questionnaire)
All interventions are rated as > 70% acceptable | 6 months
  Acceptability ratings (%); qualitative assessments; reasons for drop-outs; treatment-specific preference ratings (pre-and post-intervention)
Credibility of each component of the interprofessional intervention programme is assessed as >70% positive | 6 months
  Ratings (%) for treatment-specific expectations of benefit
Relationship between dose of nursing and response to the programme is measured | 6 months
  Amount (number), frequency ( x/day/week, intensity (+/++/+++) and duration (minutes)

SECONDARY OUTCOMES:
Study displays clinical relevance | 6 months
  How participants perceive the intervention programme (patient-reported outcomes), PROMS (51) (self-reporting closed questionnaire). Identify what is relevant for participants (such as quality of life or remaining at home) (=open question in PRO). Enables a choice of which final outcomes from the pilot study will go into the intervention (> 70%).
Cognitive function | 6 months
  Unit of measure: score from 0 to 28 Score from 0 to 28 of the Six-item Cognitive Impairment Test (6-CIT)
Multidimensional frailty | 6 months
  Score from 0 to 15 of the Tilburg Frailty Indicator (TFI)
Medication-related problems risk | 6 months
  Score from 0 to 17 of the domestic risk tool

CONTACTS AND LOCATIONS:
Overall Officials: Henk Verloo, PhD, Principal Investigator — HES-SO Valais-Wallis

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Pellegrin KL, Lee E, Uyeno R, Ayson C, Goo R. Potentially preventable medication-related hospitalizations: A clinical pharmacist approach to assessment, categorization, and quality improvement. J Am Pharm Assoc (2003). 2017 Nov-Dec;57(6):711-716. doi: 10.1016/j.japh.2017.06.019. Epub 2017 Aug 16. PMID 28823545
- [Background] Mekonnen AB, McLachlan AJ, Brien JA. Effectiveness of pharmacist-led medication reconciliation programmes on clinical outcomes at hospital transitions: a systematic review and meta-analysis. BMJ Open. 2016 Feb 23;6(2):e010003. doi: 10.1136/bmjopen-2015-010003. PMID 26908524
- [Background] Beuscart JB, Pelayo S, Robert L, Thevelin S, Marien S, Dalleur O. Medication review and reconciliation in older adults. Eur Geriatr Med. 2021 Jun;12(3):499-507. doi: 10.1007/s41999-021-00449-9. Epub 2021 Feb 13. PMID 33583002
- [Background] O'Mahony D, O'Sullivan D, Byrne S, O'Connor MN, Ryan C, Gallagher P. STOPP/START criteria for potentially inappropriate prescribing in older people: version 2. Age Ageing. 2015 Mar;44(2):213-8. doi: 10.1093/ageing/afu145. Epub 2014 Oct 16. PMID 25324330
- [Background] American Geriatrics Society 2012 Beers Criteria Update Expert Panel. American Geriatrics Society updated Beers Criteria for potentially inappropriate medication use in older adults. J Am Geriatr Soc. 2012 Apr;60(4):616-31. doi: 10.1111/j.1532-5415.2012.03923.x. Epub 2012 Feb 29. PMID 22376048
- [Background] Pereira F, von Gunten A, Rosselet Amoussou J, De Giorgi Salamun I, Martins MM, Verloo H. Polypharmacy Among Home-Dwelling Older Adults: The Urgent Need for an Evidence-Based Medication Management Model. Patient Prefer Adherence. 2019 Dec 16;13:2137-2143. doi: 10.2147/PPA.S232575. eCollection 2019. PMID 31908421
- [Background] Verloo H, Chiolero A, Kiszio B, Kampel T, Santschi V. Nurse interventions to improve medication adherence among discharged older adults: a systematic review. Age Ageing. 2017 Sep 1;46(5):747-754. doi: 10.1093/ageing/afx076. PMID 28510645
- [Background] Knight DA, Thompson D, Mathie E, Dickinson A. 'Seamless care? Just a list would have helped!' Older people and their carer's experiences of support with medication on discharge home from hospital. Health Expect. 2013 Sep;16(3):277-91. doi: 10.1111/j.1369-7625.2011.00714.x. Epub 2011 Aug 12. PMID 21838834
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Weldring T, Smith SM. Patient-Reported Outcomes (PROs) and Patient-Reported Outcome Measures (PROMs). Health Serv Insights. 2013 Aug 4;6:61-8. doi: 10.4137/HSI.S11093. eCollection 2013. PMID 25114561
- [Background] Kwan YH, Weng SD, Loh DHF, Phang JK, Oo LJY, Blalock DV, Chew EH, Yap KZ, Tan CYK, Yoon S, Fong W, Ostbye T, Low LL, Bosworth HB, Thumboo J. Measurement Properties of Existing Patient-Reported Outcome Measures on Medication Adherence: Systematic Review. J Med Internet Res. 2020 Oct 9;22(10):e19179. doi: 10.2196/19179. PMID 33034566
- [Background] Beuscart JB, Knol W, Cullinan S, Schneider C, Dalleur O, Boland B, Thevelin S, Jansen PAF, O'Mahony D, Rodondi N, Spinewine A. International core outcome set for clinical trials of medication review in multi-morbid older patients with polypharmacy. BMC Med. 2018 Feb 13;16(1):21. doi: 10.1186/s12916-018-1007-9. PMID 29433501
- [Background] O'Sullivan D, O'Regan NA, Timmons S. Validity and Reliability of the 6-Item Cognitive Impairment Test for Screening Cognitive Impairment: A Review. Dement Geriatr Cogn Disord. 2016;42(1-2):42-9. doi: 10.1159/000448241. Epub 2016 Aug 19. PMID 27537241
- [Background] Gobbens RJ, Boersma P, Uchmanowicz I, Santiago LM. The Tilburg Frailty Indicator (TFI): New Evidence for Its Validity. Clin Interv Aging. 2020 Feb 21;15:265-274. doi: 10.2147/CIA.S243233. eCollection 2020. PMID 32110005
- [Background] Katzman R, Brown T, Fuld P, Peck A, Schechter R, Schimmel H. Validation of a short Orientation-Memory-Concentration Test of cognitive impairment. Am J Psychiatry. 1983 Jun;140(6):734-9. doi: 10.1176/ajp.140.6.734. PMID 6846631
- [Background] Gobbens RJ, van Assen MA, Luijkx KG, Wijnen-Sponselee MT, Schols JM. The Tilburg Frailty Indicator: psychometric properties. J Am Med Dir Assoc. 2010 Jun;11(5):344-55. doi: 10.1016/j.jamda.2009.11.003. Epub 2010 May 8. PMID 20511102
- [Background] Deshpande PR, Rajan S, Sudeepthi BL, Abdul Nazir CP. Patient-reported outcomes: A new era in clinical research. Perspect Clin Res. 2011 Oct;2(4):137-44. doi: 10.4103/2229-3485.86879. PMID 22145124
- [Background] Male L, Noble A, Atkinson J, Marson T. Measuring patient experience: a systematic review to evaluate psychometric properties of patient reported experience measures (PREMs) for emergency care service provision. Int J Qual Health Care. 2017 Jun 1;29(3):314-326. doi: 10.1093/intqhc/mzx027. PMID 28339923